CLINICAL TRIAL: NCT01299363
Title: Vaginal Dilators for Prevention of De Novo Dyspareunia After Prolapse Surgery: A Randomized Controlled Trial
Brief Title: Dilators for Dyspareunia Prevention
Acronym: DDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: American College of Obstetricians and Gynecologists (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010-229
Record Dates: First submitted 2011-02-14; First posted 2011-02-18 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2015-04

CONDITIONS: Post-operative Dyspareunia
Keywords: Prolapse; Pain with intercourse; Dyspareunia; Post operative pain
MeSH Terms: conditions — Prolapse; Dyspareunia; Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- No dilator use (No Intervention)
- Dilator use (Active Comparator): Women randomized to vaginal dilators will be given instructions to perform softening exercises from postoperative weeks 4 to 8
  Interventions: Behavioral: Dilator use

INTERVENTIONS:
Behavioral: Dilator use — Women randomized to vaginal dilators will be given instructions to perform exercises with vaginal dilators from postoperative weeks 4 to 8
  Arms: Dilator use

SUMMARY:
This is a randomized clinical trial comparing rates of de novo dyspareunia in women with and without vaginal dilator use following surgery for pelvic organ prolapse with traditional posterior repair. Our hypothesis is daily use of vaginal dilators from post-op week 4 through week 8 after posterior repair will reduce the rate of de novo dyspareunia.

ELIGIBILITY:
Inclusion Criteria:

* Women who undergo pelvic organ prolapse surgery with a posterior repair
* Age ≥18 years
* Sexually active with heterosexual vaginal intercourse
* English speaking
* Available for 6 month follow up
* Able to complete study questionnaires
* Able to use dilators

Exclusion Criteria:

* Significant baseline dyspareunia
* Pregnancy by self-report or positive pregnancy test
* Prior pelvic radiation therapy
* Active pelvic infection, herpes, candidiasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
To compare rates of de novo dyspareunia in women with and without vaginal dilator use following surgery for pelvic organ prolapse with posterior repair (colporrhaphy). | 6 months

SECONDARY OUTCOMES:
Sexual function | 6 month
  Change in sexual function after vaginal reconstructive surgery with or without vaginal dilator use as assessed by FSFI and PISQ-12
Physical exam | 6 months
  Change in vaginal caliber and POP Q measurements 3 and 6 months after vaginal reconstructive surgery and its relation to sexual function scores and rates of dyspareunia.

CONTACTS AND LOCATIONS:
Locations (1):
- Washington Hospital Center, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Antosh DD, Gutman RE, Park AJ, Sokol AI, Peterson JL, Kingsberg SA, Iglesia CB. Vaginal dilators for prevention of dyspareunia after prolapse surgery: a randomized controlled trial. Obstet Gynecol. 2013 Jun;121(6):1273-1280. doi: 10.1097/AOG.0b013e3182932ce2. PMID 23812462